CLINICAL TRIAL: NCT01069081
Title: Phase II Study of Docetaxel and Cisplatin Chemotherapy Versus Docetaxel and Cisplatin Chemotherapy Combined With High Dose Proton Pump Inhibitor in Metastatic Breast Cancer
Brief Title: Docetaxel and Cisplatin Chemotherapy With or Without High Dose Proton Pump Inhibitor in Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Istituto Superiore di Sanità (Other)
Responsible Party: Principal Investigator, Xichun Hu, Dr, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fudan BR2010-01
Record Dates: First submitted 2010-02-10; First posted 2010-02-17 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Breast Cancer; Metastasis, Neoplasm
Keywords: Metastasis Breast Cancer; Proton Pump Inhibitor; Chemotherapy; Phase II study; TTP
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Docetaxel; Cisplatin; Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- arm A (Active Comparator): docetaxel and cisplatin chemotherapy
  Interventions: Drug: Arm A
- arm B (Experimental): docetaxel and cisplatin chemotherapy combined with PPI 160mg per day.
  Interventions: Drug: Arm B
- arm C (Experimental): docetaxel and cisplatin chemotherapy combined with PPI 200mg per day.
  Interventions: Drug: Arm C

INTERVENTIONS:
Drug: Arm C — Docetaxel and cisplatin chemotherapy combined with high dose PPI. Docetaxel 75mg/m2 intravenous d1, cisplatin 75mg/m2 intravenous d1,repeated every 3 weeks.Each patient is designed to receive no more than 6 cycles of chemotherapy.PPI 200mg p.o. d1-3 every week for 66 weeks.
  Other Names: docetaxel; cisplatin; esomeprazole
  Arms: arm C
Drug: Arm B — Docetaxel and cisplatin chemotherapy combined with lower dose PPI. Docetaxel 75mg/m2 intravenous d1, cisplatin 75mg/m2 intravenous d1,repeated every 3 weeks.Each patient is designed to receive no more than 6 cycles of chemotherapy.PPI 160mg p.o. d1-3 every week for 66 weeks.
  Other Names: Docetaxel; cisplatin; esomeprazole
  Arms: arm B
Drug: Arm A — Docetaxel and cisplatin chemotherapy. Docetaxel 75mg/m2 intravenous d1, cisplatin 75mg/m2 intravenous d1,repeated every 3 weeks.Each patient is designed to receive no more than 6 cycles of chemotherapy.
  Other Names: Docetaxel; Cisplatin
  Arms: arm A

SUMMARY:
The objectives of this study are to evaluate the efficacy and tolerability of high dose proton pump inhibitor combined with chemotherapy in metastatic breast cancer.

DETAILED DESCRIPTION:
High dose proton pump inhibitor (PPI) has been proved beneficial and it improved efficacy when combined with chemotherapy in preclinical and clinical trials.This study was designed to explore whether adding a proton pump inhibitor into docetaxel and cisplatin chemotherapy improves efficacy and does not affect tolerability in metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Female, ≥ 18 years.
* Histologically confirmed invasive breast cancer.
* Metastatic breast cancer.
* Karnofsky Performance Status ≥60.
* Life expectancy of more than 3 months.
* Subject must have adequate organ function.
* Normal laboratory values: hemoglobin > 80g/dl, neutrophils > 2.0×10^9/L, platelets > 80×10^9/L, serum creatinine < upper limit of normal (ULN), serum bilirubin < ULN, ALT and AST < 2.5×ULN, AKP < 5×ULN.
* Negative serum pregnancy test for women with childbearing potential.
* Good conditions for infusion and willing to have phlebotomy throughout whole study.
* Have ceased anti-tumor treatments including endocrinotherapy and bio-targeted therapy for more than 28 days.
* Have at least one target lesion according to the Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
* No prior use of docetaxel or has used docetaxel in adjuvant/neo-adjuvant chemotherapy and has a relapse free survival of at least 12 months.

Exclusion Criteria:

* Pregnant or lactating females.
* History of other malignancy. However, subjects who have been disease-free for 5 years, or subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible.
* Concurrent disease or condition that would make the subject inappropriate for study participation, or any serious medical disorder that would interfere with the subject's safety.
* Active or uncontrolled infection.
* Known history of uncontrolled or symptomatic angina, arrhythmias, or congestive heart failure.
* Concomitant with brain metastases.
* Have received chemotherapy after metastasis.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2009-08; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Time to progression | six weeks

SECONDARY OUTCOMES:
Time to treatment failure,Objective response,Overall survival,Safety | six weeks

CONTACTS AND LOCATIONS:
Overall Officials: XiChun Hu, MD,Ph. D, Principal Investigator — Fudan University; Antonio Chiesi, Principal Investigator — Istituto Superiore di Sanità; Stefano Fais, MD PHD, Study Director — Istituto Superiore di Sanità
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Wang BY, Zhang J, Wang JL, Sun S, Wang ZH, Wang LP, Zhang QL, Lv FF, Cao EY, Shao ZM, Fais S, Hu XC. Intermittent high dose proton pump inhibitor enhances the antitumor effects of chemotherapy in metastatic breast cancer. J Exp Clin Cancer Res. 2015 Aug 22;34(1):85. doi: 10.1186/s13046-015-0194-x. PMID 26297142